CLINICAL TRIAL: NCT01602679
Title: Acute Effects of Progesterone on LH Pulses During the Follicular Phase
Brief Title: Acute Effects of Progesterone on LH Pulses During the Follicular Phase (CRM006)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Interim analysis suggested futility.
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chris McCartney, Associate Professor of Medicine, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 16085; R01HD058671 (NIH)
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Female Reproductive Physiology
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- micronized progesterone, then placebo (Experimental): Participants first received oral micronized progesterone (100 mg p.o.) suspension. After a washout period of approximately 20 days, they then received placebo (matching oral micronized progesterone suspension).
  Interventions: Drug: oral micronized progesterone suspension; Drug: Placebo
- Placebo, then micronized progesterone (Placebo Comparator): Participants first received placebo. After a washout period of approximately 20 days, they then received oral micronized progesterone syrup (100 mg p.o.)Placebo contains only inert ingredients and is not expected to exert any direct physiological effects
  Interventions: Drug: oral micronized progesterone suspension; Drug: Placebo

INTERVENTIONS:
Drug: oral micronized progesterone suspension — oral micronized progesterone (100 mg p.o.) suspension
  Other Names: Progesterone
Drug: Placebo — Placebo contains only inert ingredients and is not expected to exert any direct physiological effects

SUMMARY:
The rapidity with which progesterone slows LH (and by inference GnRH) pulse frequency in women is unclear. The investigators hypothesize that progesterone slows LH pulse frequency within 10 hours. The investigators propose to assess this further with a randomized, cross-over, placebo-controlled study. Regularly cycling women without hyperandrogenism will be admitted to the Clinical Research Unit on cycle day 5-9 (mid-follicular phase) for a 10 hour frequent sampling study to observe LH, FSH, estradiol, progesterone, and testosterone. Either oral micronized progesterone suspension or placebo will be administered at 0900 h. During a subsequent menstrual cycle, subjects will undergo another study identical to the first except that oral progesterone will be exchanged for placebo or vice versa in accordance with a crossover design.

DETAILED DESCRIPTION:
The rapidity with which progesterone slows LH (and by inference GnRH) pulse frequency in women is unclear. The investigators hypothesize that progesterone slows LH pulse frequency within 10 hours. The investigators propose to assess this further with a randomized, cross-over, placebo-controlled study. Regularly cycling women without hyperandrogenism will be admitted to the Clinical Research Unit on cycle day 5-9 (mid-follicular phase) for a frequent sampling study. Beginning at 0900 h, blood for LH, FSH, estradiol, progesterone, and testosterone will be obtained over a 10-hour period. Either oral micronized progesterone (100 mg p.o.) suspension or placebo will be administered at 0900 h. During a subsequent menstrual cycle, subjects will undergo another study identical to the first except that oral progesterone will be exchanged for placebo or vice versa in accordance with a crossover design. The primary endpoint of interest is LH pulse frequency; the investigators will compare LH pulse frequency after progesterone administration to LH pulse frequency after placebo administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be healthy women with regular menstrual cycles and no evidence of hyperandrogenism.
* Subjects will be 18-30 years old; the investigators use a cutoff age of 30 years because age-related alterations in the hypothalamic-pituitary-ovarian axis is uncommon before age 30 years.
* Subjects will be willing to strictly avoid pregnancy (using non-hormonal methods) during the time of study and must be willing and able to provide informed consent.

Exclusion Criteria:

* Pregnancy
* Lactation
* History of allergy to progesterone
* BMI < 18 kg/m2 or > 30 kg/m2 (underweight and obesity can affect hypothalamic-pituitary-ovarian function)
* Excessive exercise, defined as routine and current engagement in either (a) moderate exercise (e.g., brisk walking) exceeding 14 hours per week or (a) vigorous exercise exceeding 7 hours a week.
* Clinical hyperandrogenism (primarily hirsutism)
* Abnormally elevated free testosterone or DHEAS concentration
* A previous diagnosis of diabetes, a fasting glucose ≥ 126 mg/dl
* Abnormal TSH (subjects with adequately treated hypothyroidism, reflected by normal TSH values, will not be excluded; or, for a new diagnosis of hypothyroidism, further study will at the least be delayed pending appropriate treatment) (confirmed on repeat)
* Abnormal prolactin (confirmed on repeat)
* Evidence of Cushing's syndrome by history or physical exam
* History of venous thromboembolism, breast/ovarian/endometrial cancer
* The investigators will exclude women with any other cancer diagnosis and/or treatment (with the exception of basal cell or squamous skin carcinoma) unless they have remained clinically disease free (based on appropriate surveillance) for five years.
* Women with anemia (hematocrit < 36% and hemoglobin level < 12 g/dl) will be treated with iron for a maximum of 2 sequential months before the 1st admission and/or before the 2nd admission. If they remain anemic after 2 sequential months of ferrous gluconate (325 mg bid), they will then be excluded from further participation in the study.
* Women with a significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure; known or suspected coronary atherosclerosis; asthma requiring systemic intermittent corticosteroids; etc.) will be excluded.
* Women with liver enzymes, alkaline phosphatase, or bilirubin > 1.5 times upper limit of normal (confirmed on repeat) will be excluded, with the exception that mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome.
* Abnormal sodium or potassium concentrations (confirmed on repeat); bicarbonate concentrations <20 or >30 (confirmed on repeat)
* Women with abnormal renal function (i.e., serum creatinine > 1.4) will be excluded (confirmed on repeat)
* Due to the amount of blood being drawn in the study, subjects with body weight < 110 pounds will be excluded from the study
* Being a study of the acute effects of progesterone on the hypothalamic-pituitary unit, subjects must not take hormonal medications (e.g., oral contraceptives) or other medications known to affect the reproductive axis for 60 days prior to the study and during the study.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. McCartney, MD, Principal Investigator — University of Virginia
Locations (1):
- Center for Research in Reproduction, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not have current plans to share IPD

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 subjects enrolled in this study. 5 subjects completed screening procedures only (these 5 subjects were withdrawn from study prior to being assigned to an arm of intervention).
Groups:
- Oral Micronized Progesterone Suspension, Then Placebo: Participants first received oral micronized progesterone (100 mg p.o.) suspension. After a washout period of approximately 20 days, they then received placebo.
  oral micronized progesterone suspension: oral micronized progesterone (100 mg p.o.) suspension
- Placebo, Then Oral Micronized Progesterone Suspension: Participants first received Placebo. After a washout period of approximately 20 days, they then received oral micronized progesterone suspension. Placebo contains only inert ingredients and is not expected to exert any direct physiological effects
  Placebo: Placebo contains only inert ingredients and is not expected to exert any direct physiological effects
Period: Overall Study
Arm/Group | Oral Micronized Progesterone Suspension, Then Placebo | Placebo, Then Oral Micronized Progesterone Suspension
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Oral Micronized Progesterone Suspension, Then Placebo: Participants first received oral micronized progesterone (100 mg p.o.) suspension. After a washout period of approximately 20 days, they then received Placebo.
  oral micronized progesterone suspension: oral micronized progesterone (100 mg p.o.) suspension Placebo: Placebo contains only inert ingredients and is not expected to exert any direct physiological effects
- Placebo, Then Oral Micronized Progesterone Suspension: Participants first received Placebo. After a washout period of approximately 20 days, they then received oral micronized progesterone suspension. Placebo contains only inert ingredients and is not expected to exert any direct physiological effects
  Placebo: Placebo contains only inert ingredients and is not expected to exert any direct physiological effects oral micronized progesterone suspension: oral micronized progesterone (100 mg p.o.) suspension
- Total: Total of all reporting groups
Arm/Group | Oral Micronized Progesterone Suspension, Then Placebo | Placebo, Then Oral Micronized Progesterone Suspension | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of LH Pulses Per Hour
Description: The primary endpoint is the change in the number of LH pulses per hour (over 10 h), comparing (a) number of LH pulses at baseline to (b) number of LH pulses immediately after progesterone or placebo administration
Time Frame: 10 hours following administration of micronized progesterone or placebo
Measure: Mean (Standard Deviation); unit: pulses/h
Arm/Group | Oral Micronized Progesterone Suspension | Placebo
Number analyzed (Participants) | 7 | 7
pulses/h | 0.77 (0.28) | 0.79 (0.35)

2. Secondary Outcome: Change in Mean LH
Description: This secondary endpoint is the change of the mean LH (over 10 h), comparing (a) mean LH at baseline to (b) mean LH immediately after progesterone or placebo administration
Time Frame: 10 hours following administration of micronized progesterone or placebo
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Oral Micronized Progesterone Suspension | Placebo
Number analyzed (Participants) | 7 | 7
IU/L | 5.8 (2.2) | 4.6 (2.3)

3. Secondary Outcome: Change in Mean LH Amplitude
Description: This secondary endpoint is the change in the mean LH amplitude (over 10 h), comparing (a) mean LH amplitude at baseline to (b) mean LH amplitude immediately after progesterone or placebo administration
Time Frame: 10 hours following administration of micronized progesterone or placebo
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Oral Micronized Progesterone Suspension | Placebo
Number analyzed (Participants) | 7 | 7
IU/L | 4.3 (2.8) | 3.6 (2.8)

ADVERSE EVENTS:
Time Frame: From start of study procedures until end of study participation, up to 6 months
Groups:
- Oral Micronized Progesterone Suspension: Oral micronized progesterone (100 mg) suspension
Arm/Group | Oral Micronized Progesterone Suspension | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/4 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Micronized Progesterone Suspension (N=4) | Placebo (N=3)
Irregular Menstrual Bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Temporary spotting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT01602679/Prot_SAP_000.pdf